CLINICAL TRIAL: NCT00973388
Title: A Double-blind, Double-dummy, Randomized, Placebo- and Active-controlled, Four-period Crossover Trial to Evaluate the Effect of Telaprevir (TVR) on the QT/QTc Interval in Healthy Subjects
Brief Title: VX-950-TiDP24-C136 - A Trial to Evaluate the Effect of Telaprevir (TVR) on the Results of Electrocardiograms (Electric Recording of the Heart) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR016417
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C
Keywords: VX-950-TiDP24-C136; VX-950-C136; VX-950; HEPATITIS; Telaprevir; Moxifloxacin; ECG; QT; QTc
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — telaprevir; Moxifloxacin

INTERVENTIONS:
Drug: Telaprevir; Moxifloxacin; Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of telaprevir on the results of electrocardiograms in healthy volunteers. An electrocardiogram is an electric recording of the heart. Telaprevir is being investigated for the treatment of chronic hepatitis C virus infection.

DETAILED DESCRIPTION:
This is a Phase I, double-blind, double-dummy, randomized, placebo- and active-controlled, 4-period crossover trial. This means the study doctor nor yourself know in which treatment session you will receive which active medication or matching placebo. Every participant will receive each treatment in turn. The order in which you receive the treatment sessions is determined by chance, like tossing a coin. The purpose of the study is to evaluate the effect of telaprevir (TVR) on the results of electrocardiograms (electric recording of the heart). Two dose regimens of TVR will be tested, i.e. 750 mg every 8 hours (the dose that will be given to patients) and 1875 mg every 8 hours (a dose higher than the one that will be given to patients), administered for 4 days, with an additional morning dose on Day 5. A single dose of 400 mg moxifloxacin will be used as a positive control to assess trial sensitivity. The trial population will consist of 44 healthy volunteers. Treatment A will consist of TVR 750 mg every 8 hours on Days 1-4 + single 750 mg morning dose on Day 5 (2 active TVR tablets + 3 TVR placebo tablets every 8 hours on Days 1 to 4 with a single morning dose on Day 5, and a single morning dose of moxifloxacin placebo on Day 5). Treatment B will consist of TVR 1875 mg every 8 hours on Days 1 to 4 + single 1875 mg morning dose on Day 5 (5 active TVR tablets every 8 hours on Days 1 to 4 with a single morning dose on Day 5, and a single morning dose of moxifloxacin placebo on Day 5). Treatment C will consist of a single dose of 400 mg moxifloxacin (5 TVR placebo tablets every 8 hours on Days 1 to 4 with a single morning dose on Day 5, and a single morning dose of active moxifloxacin on Day 5). Treatment D will consist of placebo (5 TVR placebo tablets every 8 hours on Days 1 to 4 with a single morning dose on Day 5, and a single morning dose of moxifloxacin placebo on Day 5).There will be a washout period of 8 days between subsequent treatment sessions. Electrocardiograms (ECGs) will be recorded continuously for 24 hours by Holter monitoring (small electrodes will be attached to your chest and connected to a small device to record your heart rhythm over a 24-hour period) on the day before intake of study medication starts and on Day 5 of all treatment sessions. In addition, for safety monitoring, separate ECGs will be performed at predefined time points. Samples to access pharmacokinetics (how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body) of TVR and moxifloxacin will be collected on the day before intake of medication starts and day 5 of all treatment sessions, as well as predose on Days 2, 3 and 4 of all treatment sessions. Safety and tolerability will be evaluated throughout the trial by evaluating results of blood- and urine analysis, vital signs, physical examinations, alcohol breath tests and by assessing how you are feeling. In every treatment session, participants will receive 5 oral tablets of 375 mg TVR or placebo every 8 hours on Days 1 to 4 with a single morning dose on Day 5, and a single oral morning dose of 400 mg moxifloxacin or placebo on Day 5. In between treatment sessions, there will be a wash-out period of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking for at least 6 months prior to screening
* A body mass index (BMI, weight in kg divided by the square of height in meters) of 18 to30 kg/m2, extremes included
* Otherwise healthy on the basis of a physical examination, medical history, electrocardiogram, vital signs and the results of laboratory tests and a urinalysis carried out at screening

Exclusion Criteria:

* Consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week from 14 days before the first intake of study medication and of an average of more than five 240-mL servings of coffee or other caffeinated beverage (e.g. tea, cola) per day from screening onwards
* A history of drug or alcohol abuse or addiction within 2 years prior to dosing, or a positive test for alcohol or drugs during the screening period
* Participation in a clinical study involving administration of an investigational drug within 2 months or 5 half lives (whichever is longer) prior to the screening visit
* Donation of any blood or having had a significant loss of blood within 3 months, or donation of more than 1 unit of plasma within 7 days before the first dose of study drug
* Male patients with female partners who are planning to become pregnant during the study or within 90 days of the last dose of study medication and female patients of childbearing potential who are pregnant or planning to become pregnant within 90 days of the completion of the study, who are not using adequate contraception, or who are breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of administration of TVR 750 mg every 8 hours and 1875 mg every 8 hours, both at steady-state, versus placebo on the QT and QTc interval (heart activity) in healthy volunteers. | For each dosing period, QT/QTc data will be recorded continuously for 24 hours by 12-lead Holter monitoring on Day-1 and Day 5. Time-matched triplicate ECGs at predose, and at 1, 2, 3, 4, 5, 6, 8 and 24 hour time points will be extracted.

SECONDARY OUTCOMES:
Trial sensitivity will be evaluated (i.e., the effect of a positive control, a single 400 mg dose of moxifloxacin, on the QT/QTc interval). | In treatment session C, QT/QTc data will be recorded continuously for 24 hours by 12-lead Holter monitoring on Day-1 and Day 5. Time-matched triplicate ECGs at predose, and at 1, 2, 3, 4, 5, 6, 8 and 24 hour time points will be extracted.
The effect of 2 different regimens of TVR on non-QT interval electrocardiogram (ECG) parameters (RR interval, HR, PR interval, and QRS interval) will be evaluated. | In treatment session A and B, QT/QTc data will be recorded continuously for 24 hours by 12-lead Holter monitoring on Day-1 and Day 5. Time-matched triplicate ECGs at predose, and at 1, 2, 3, 4, 5, 6, 8 and 24 hour time points will be extracted.
The pharmacokinetics of 2 dose regimens of TVR, 750 mg every 8 hours and 1875 mg every 8 hours, at steady-state will be evaluated. | Samples to access pharmacokinetics of TVR will be collected on Days -1 and 5 of each treatment session (8 times sampling in a period of 9 hours), as well as predose on Days 2, 3 and 4 of each treatment session.
The concentration-effect relationship for QT/QTc for TVR will be explored. | In each treatment session, QT/QTc data will be recorded continuously for 24 hours by 12-lead Holter monitoring on Day-1 and Day 5. Time-matched triplicate ECGs at predose, and at 1, 2, 3, 4, 5, 6, 8 and 24 hour time points will be extracted.
The short-term safety and tolerability of 2 dose regimens of TVR, 750 mg and 1875 mg every 8 hours will be evaluated. | Safety will be assessed from screening until the last trial related visit (approximately 15 weeks). Tolerability will be evaluated from the first dosing in the first treatment session until the last trial related visit (approximately 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA